CLINICAL TRIAL: NCT00168194
Title: Cellular Immune Responses to Hepatitis B Virus (HBV)- Longitudinal Follow up and Natural History
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Hoy, Professor Jennifer Hoy, The Alfred
Other Study IDs: 235/04
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Hepatitis B; HIV Infections
Keywords: HIV
MeSH Terms: conditions — Hepatitis B; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
It remains unclear why some individuals are able to clear HBV from their bodies while in others HBV is a persistent infection. We plan to investigate this process by collecting blood and analysing how the patient's white blood cells respond to different pieces of the HBV virus. We will use new tools that can precisely tell us which component of the immune response may be different in individuals who are chronically infected with HBV and also in individuals who are also infected with HIV.

The primary aims are therefore:

1. To characterize HBV-specific T cell responses in HBV chronic carriers, and identify novel immunogenic regions in both HLA-A2+ and non-HLA-A2+ individuals.
2. To determine the effect of HIV infection on HBV-specific T-cell responses

ELIGIBILITY:
Inclusion Criteria:

There are two groups of patients in this study. Group A mono-infected with Hepatitis B, and those with co-infection HBV/HIV.

Group A inclusion criteria: (also split into 6 recruiting groups)

* Acute hepatitis B
* Chronic hepatitis B, HBV DNA+ve , normal ALT , HBeAg +ve
* Chronic hepatitis B, HBV DNA +ve , normal ALT, HBeAg -ve
* Chronic hepatitis , HBV DNA +ve, increased ALT, no HBV treatment B, HBeAg +ve
* Chronic hepatitis B, HBV DNA +ve , increased ALT, no HBV treatment B, HBeAg -ve
* Chronic hepatitis B, undergoing 'flare' of hepatitis

Group B inclusion criteria:

* To be HIV/HBV co-infected

All patients:

* To be over 18 years

Exclusion Criteria:

* Those who do not fit the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV and hepatitis B co-infection
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2004-12; Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lewin, Professor, Principal Investigator — Burnet Institute, Melbourne
Locations (1):
- The Alfred Hospital, Commercial Road, Melbourne, Victoria, Australia